



| NCT Number: NCT04370691 |
|--------------------------------------------------------|
| JETi Registry |
| JET Enhanced Thrombectomy intervention (JETi) Registry |
| Study Document No: |
| Version |
| Date: 17-Aug-2024 |

Sponsor: Abbott



## **Statistical Analysis Plan**

CIP Number: JETi Registry

<u>JET Enhanced Thrombectomy intervention (JETi)</u>
Registry

**Statistical Analysis Plan (SAP)** 



## **Statistical Analysis Plan**

## **TABLE OF CONTENTS**

| SYNOPSIS OF STUDY DESIGN4 |
|--------------------------------------------------------|
| 1.1 Purpose of the Statistical Analysis Plan |
| 1.2 Clinical Investigation Objectives |
| 1.3 Clinical Investigation Design |
| 1.4 Endpoints4 |
| 1.4.1 Primary Endpoints4 |
| 1.4.1.1 Arterial Subjects4 |
| 1.4.1.2 Venous Subjects5 |
| 1.4.2 Descriptive Endpoint(s) |
| 1.4.2.1 All Subjects5 |
| 1.4.2.2 Arterial Subjects6 |
| 1.4.2.3 Venous Subjects |
| 2.0 ANALYSIS CONSIDERATIONS |
| 2.1 Analysis Populations8 |
| 2.2 Statistical Methods8 |
| 2.2.1 Descriptive Statistics for Continuous Variables |
| 2.2.2 Descriptive Statistics for Categorical Variables |
| 2.3 Endpoint Analysis |
| 2.3.1 Primary Endpoint(s)9 |
| 2.3.1.1 Arterial Subjects9 |
| 2.3.1.2 Venous Subjects 9 |
| 2.3.2 Descriptive Endpoint(s) Analyses |
| 2.6 Timing of Analysis |
| 2.9 Handling of Missing Data11 |
| 2.10 Poolability Issue 12 |
| 3.0 DESCRIPTIVE ENDPOINTS AND ADDITIONAL DATA |



## **Statistical Analysis Plan**

| 3.1 | Baseline and Demographic Characteristics | . 12 |
|-----|------------------------------------------|------|
| 3.2 | Adverse Events | . 12 |
| 3.3 | Subject Early Termination | . 13 |
| 3.4 | Protocol Deviation | . 13 |
| 4.0 | DOCUMENTATION AND OHER CONSIDERATIONS | . 13 |
| 5.0 | ACRONYMS AND ABBREVIATIONS | . 14 |
| 6.0 | REFERENCES | . 15 |
| 7 0 | APPENDICES | 15 |



### Statistical Analysis Plan

### 1.0 SYNOPSIS OF STUDY DESIGN

#### 1.1 Purpose of the Statistical Analysis Plan

| This statistical analysis plan (SAP) is intended to p | provide a detailed and comprehensive description of |
|---|---|
| the planned methodology and analysis to be used | for the JETi Registry clinical |
| investigation. This plan is based on the | Clinical Investigation Plan. |

#### 1.2 Clinical Investigation Objectives

The objective of the JETi Registry is to collect real-world data on the safety, performance, and clinical benefits of the JETi System for the treatment of thrombosis in the peripheral vasculature.

#### 1.3 Clinical Investigation Design

The JETi Registry is a prospective, single-arm, multicenter study to collect real-world data on the safety, performance, and clinical benefits of the JETi System for the treatment of acute and subacute thrombosis in the peripheral vasculature. This is a post-market study and will register approximately 280 subjects at approximately 30 centers globally. Subjects participating in this registry will be followed through their 12-month follow up visit.

After JETi procedure,

subjects will be evaluated at discharge, 30 days, and 12 months.

#### 1.4 Endpoints

#### 1.4.1 Primary Endpoints

#### 1.4.1.1 Arterial Subjects

For subjects treated for arterial or arteriovenous thrombosis, the primary endpoints are:

Clot removal grade for each JETi-treated target vessel(s) from pre-JETi angiogram to post-JETi
angiogram (post-JETi thrombectomy and prior to any adjunctive therapies to treat underlying
culprit lesions) per the grades in Table 1 (vessel basis). The independent imaging core laboratory
will be responsible for assessing this endpoint.

Table 1. Clot Removal Grade

| Grade I | < 50% reduction |
|-----------|---------------------|
| Grade II | 50 - <95% reduction |
| Grade III | 95 – 100% reduction |

Composite of JETi-related major adverse events (MAEs), defined as the following JETi-related
events: device-related death, major amputation of the treated limb (arterial subjects only), or
major bleeding up to 30 days post-JETi procedure and as adjudicated by a clinical events
committee (CEC) (subject basis).



## Statistical Analysis Plan

#### 1.4.1.2 Venous Subjects

For subjects treated for lower extremity DVT, the primary endpoints are

Percent of treated vessel(s) with ≥ 75% venous thrombus reduction from pre-JETi venogram
to final venogram (post-JETi AND after any/all adjunctive therapies to treat underlying culprit
lesions) via modified Marder score. The independent imaging core laboratory will be responsible
for assessing this endpoint.

If no adjunctive therapies or devices are used after JETi, post-JETi modified Marder score is also final score.

 Composite of JETi-related major adverse events (MAEs), up to 30 days post-JETi procedure, defined as the following JETi-related events, adjudicated by a clinical event committee (CEC): (1) death, (2) symptomatic pulmonary embolism (PE), (3) major bleeding, (4) re-thrombosis of JETitreated vessel(s).



#### 1.4.2 Descriptive Endpoint(s)

#### 1.4.2.1 All Subjects

- Procedure-related death as adjudicated by a CEC.
- JETi-related AEs collected at discharge, 30 days, and 12 months follow-up, and as adjudicated by a CEC.
- Procedure-related access site complications such as hematoma, pseudoaneurysm (false aneurysm), perforation, as adjudicated by a CEC.



## Statistical Analysis Plan

• Treatment Used: The number and percentage of patients having each of the following treatments:



Quality of life (QoL) questionnaire: SF-12 at baseline, 30-day and 12-month follow-up.

#### 1.4.2.2 Arterial Subjects

- Clot removal grade for each JETi-treated target vessel from pre-JETi angiogram to final
  angiogram (post-JETi thrombectomy and after any/all adjunctive therapies and prior to removal of
  the vascular sheath) per the grades in Table 1.
- Components of the MAE including device-related death, major amputation of treated limb (arterial subjects only), and major bleeding up to 30 days post-JETi as adjudicated by a CEC.
- Ankle Brachial Index\* (ABI) of treated limb(s) at baseline and 30 days.
- Rutherford\* classification at baseline and 30 days.
   \* only applicable to subjects with lower limb arterial thrombus.
- Rate of re-thrombosis of JETi-treated vessel at 30 days, and 12 months, as assessed by investigator/physician reported.
- Patency as determined by duplex ultrasound at baseline, 30-day, and 12-month follow-up. Note that this endpoint will only apply to subjects treated for arteriovenous thrombus.
- Vessel patency: assessed by the independent imaging core laboratory using the Modified Thrombolysis in Myocardial Infarction (TIMI) classification called TIPI (Thrombo-aspiration in Peripheral Ischemia)<sup>1</sup> (Table 3) for each JETi-treated vessel, assessed using angiogram.
  - At post-JETi timepoint (post-JETi thrombectomy <u>and prior</u> to any adjunctive therapies to treat underlying culprit lesions)
  - At final timepoint (post-JETi thrombectomy <u>and after</u> any/all adjunctive therapies and prior to removal of the vascular sheath)

<sup>&</sup>lt;sup>1</sup> de Donato G, Pasqui E, Sponza M, et al. Safety and Efficacy of Vacuum Assisted Thrombo-Aspiration in Patients with Acute Lower Limb Ischaemia: The INDIAN Trial. *Eur J Vasc Endovasc Surg*. 2021;61(5):820-828. doi:10.1016/j.ejvs.2021.01.004



## **Statistical Analysis Plan**

If no adjunctive therapies or devices are used after JETi, post-JETi TIPI score is also final TIPI score.

Table 3. Thrombo-aspiration in Peripheral Ischemia (TIPI)

| Description | TIPI score |
|---|---|
| No recanalization of the thrombotic occlusion | 0 |
| Incomplete or partial recanalization of the thrombotic occlusion with no distal flow | 1 |
| Incomplete or partial recanalization of the thrombotic occlusion with any distal flow | 2 |
| Complete recanalization of the thrombotic occlusion with normal distal flow | 3 |

- Acute success, as per TIPI score (Table 3), per core lab assessment:
  - Device success: Near complete or complete recanalization of occluded vessel, defined as post-JETi TIPI 2-3.
  - Technical success: Near complete or complete recanalization of occluded vessel, defined as final TIPI 2-3, using JETi system and any other adjunctive device or procedures.
  - Procedural success: Technical success with no JETi-related MAEs within 5 days of registration or by discharge, whichever occurs first.

#### 1.4.2.3 Venous Subjects

- Percent of treated vessels with ≥75% clot reduction from pre-JETi venogram to post-JETi venogram (post-JETi thrombectomy and before any adjunctive therapies to treat underlying culprit lesions) via modified Marder score. The independent imaging core laboratory will be responsible for assessing this endpoint.
- For subjects not treated for lower extremity DVT (i,e. upper extremity DVT (UE DVT)), Clot removal grade for each JETi-treated target vessel from pre-JETi venogram to final venogram (post-JETi thrombectomy and after any/all adjunctive therapies and prior to removal of the vascular sheath) per the grades in **Table 1**.
- Components of the JETi-related MAE including up to 30 days post-JETi adjudicated by a CEC death, symptomatic pulmonary embolism (PE), major bleeding and rethrombosis of target vessel(s).
- Re-thrombosis in the JETi-treated vessel(s) at 30-day and 12-month follow up, as assessed by investigator/physician reported, and as adjudicated by CEC.
- The Villalta Post Thrombotic Syndrome (PTS) severity scale at baseline, 30-day, and 12-month follow-up. Note that this assessment will apply only to subjects with lower extremity DVT.



## **Statistical Analysis Plan**

- Edema component score from the Villalta Post Thrombotic Syndrome (PTS) severity scale at baseline, 30-day, and 12-month follow-up.
- A 7-point Likert Scale for leg pain at baseline, discharge, 30-day, and 12-month follow-up.
- Venous patency and compressibility as determined by duplex ultrasound at baseline, 30-day, and 12-month follow-up.
- Acute success,
   assessed by core laboratory:
  - Device success: Post-JETi thrombus removal grade II-III
  - occurs after JETi system and any other adjunctive device or procedures.
  - Procedural success: Technical success with no JETi-related MAEs within 5 days of registration or by discharge, whichever occurs first.

If no adjunctive therapies or devices are used after JETi, post-JETi is also final score



#### 2.0 ANALYSIS CONSIDERATIONS

### 2.1 Analysis Populations

All registered subjects will be included in the analyses. The point of registration in the Registry is when a JETi Catheter is introduced into the intended vasculature of an enrolled subject during the procedure (Day 0). A subject who is enrolled but not registered in this study will be considered as a screen failure.

Consenting up to 5 days post-JETi procedure is acceptable. In these cases, the point of registration will be the same and any procedural information will be entered post-consent, and adverse events (AEs) will be collected retrospectively from the point of registration (Day 0).

#### 2.2 Statistical Methods

#### 2.2.1 Descriptive Statistics for Continuous Variables

For continuous variables (e.g., age, BMI, etc.), results will be summarized with the numbers of observations, means, and standard deviations, with quartiles, minimums, maximums, and 95% confidence intervals, where specified.

#### 2.2.2 Descriptive Statistics for Categorical Variables





## Statistical Analysis Plan

#### 2.3 Endpoint Analysis

#### 2.3.1 Primary Endpoint(s)

#### 2.3.1.1 Arterial Subjects

For subjects treated for arterial thrombosis

all endpoints are

descriptive. There will be no hypothesis testing, and there are no statistical power considerations.

#### Primary Effectiveness Endpoint:

Clot removal grade for each JETi-treated target vessel from pre-JETi angiogram to post-JETi angiogram (post-JETi thrombectomy and prior to any adjunctive therapies to treat underlying culprit lesions) per the grades. Summary statistics (number and % of treated vessel) of clot removal grade from pre- to post-JETi thrombectomy will be summarized.

#### Primary Safety Endpoint:

Composite of JETi-related major adverse events (MAEs), defined as the following JETi-related events: device-related death, major amputation of the treated limb (arterial subjects only), or major bleeding up to 30 days post-JETi procedure and as adjudicated by a clinical events committee (CEC). It will be summarized as the number of events and the percentage of subjects with events.

#### 2.3.1.2 Venous Subjects

#### Primary Effectiveness Endpoint:

• For subjects treated for lower extremity DVT, the primary effectiveness endpoint is the percent of treated vessel(s) with ≥ 75% venous thrombus reduction from pre-JETi venogram to final venogram (post-JETi AND after any/all adjunctive therapies to treat underlying culprit lesions) via modified Marder score. If no adjunctive therapies or devices are used after JETi, post-JETi modified Marder score is also final score. This endpoint is a binary outcome defined as whether there is 75% reduction in modified Marder score from baseline at the limb level.





## **Statistical Analysis Plan**



#### **Primary Safety Endpoint:**

The primary safety endpoint is the composite of JETi-related MAEs, up to 30 days post- JETi procedure (death, symptomatic pulmonary embolism (PE), major bleeding, or re-thrombosis of JETi-treated vessel(s)) for subjects treated for lower extremity DVT and as adjudicated by a clinical events committee (CEC).

It will be summarized as the number of events and the percentage of subjects with events.



#### 2.3.2 Descriptive Endpoint(s) Analyses

All descriptive endpoints will be summarized descriptively.





## Statistical Analysis Plan

| A total of approximately 280 subjects will be registered in this Registry. |
|----------------------------------------------------------------------------|

#### 2.6 Timing of Analysis

Analysis for the primary endpoints will be performed after all registered subjects (within arterial or DVT groups) have reached their 30-day follow-up visit. Analysis for final report will be conducted after all registered subjects have completed the 12-month follow-up visit.



Analysis will be performed separately for arterial and venous subjects.

### 2.9 Handling of Missing Data

Every effort will be made to acquire all necessary data. Analysis will be based on available data with missing data excluded. Any unused or spurious data will be noted as appropriate in the final report. However, impact of missing data may be assessed in the sensitivity analysis.



## Statistical Analysis Plan

## 2.10 Poolability Issue



#### 3.0 DESCRIPTIVE ENDPOINTS AND ADDITIONAL DATA

### 3.1 Baseline and Demographic Characteristics

The following baseline and demographic variables will be summarized for all registered subjects: gender, age, ethnicity, race, medical history, etc.

#### 3.2 Adverse Events

All device-, and procedure-related adverse events and all serious adverse events will be summarized for all registered subjects in this trial in terms of the number of events, the percentage of subjects with events.





## **Statistical Analysis Plan**

#### 3.3 **Subject Early Termination**

Subject early termination reasons including deaths, withdrawals, lost-to-follow-up, etc. will be summarized at all scheduled visits.

#### 3.4 **Protocol Deviation**

Protocol deviations will be summarized for subjects in whom a protocol deviation was reported.

#### 4.0 **DOCUMENTATION AND OHER CONSIDERATIONS**

All analyses will be performed using SAS® for Windows, version 9.4 or higher.



## **Statistical Analysis Plan**

## 5.0 **ACRONYMS AND ABBREVIATIONS**

| Acronym or Abbreviation | Complete Phrase or Definition |
|-------------------------|-------------------------------------------|
| ABI | Ankle Brachial Index |
| ALI | Acute Limb Ischemia |
| AV | Arteriovenous |
| CDT | Catheter Directed Thrombolysis |
| CEC | Clinical Events Committee |
| CIP | Clinical Investigation Plan |
| DVT | Deep Vein Thrombosis |
| IVC | Inferior Vena Cava |
| MAE | Major Adverse Event |
| OUS | Outside of US |
| PE | Pulmonary Embolism |
| PG | Performance Goal |
| PTS | Post Thrombotic Syndrome |
| QOL | Quality of Life |
| SAE | Serious Adverse Event |
| SAP | Statically Analysis Plan |
| SF-12 | Short-Form Health Survey-12 |
| TIMI | Thrombolysis in Myocardial Infarction |
| TIPI | Thrombo-aspiration in Peripheral Ischemia |



## Statistical Analysis Plan

## 6.0 **REFERENCES**

2. SAS Institute Inc. 2015. SAS/STAT® 14.1 User's Guide. Cary, NC: SAS Institute Inc.

## 7.0 **APPENDICES**



## Statistical Analysis Plan

### APPENDIX A: STATISTICAL ANALYSIS PLAN REVISIONS

